CLINICAL TRIAL: NCT04478578
Title: Determining the Incidence, Causes and Outcomes of Rural Febrile Illness (RFI) in South and Southeast Asia, as Part of the South and Southeast Asian Community-based Trials Network (SEACTN). Work Package A (WP-A).
Brief Title: Incidences, Causes, and Outcomes of Febrile Illness in Rural South and Southeast Asia
Acronym: SEACTN-WP-A
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Medical Action Myanmar (Other); Shoklo Malaria Research Unit (Other); Lao-Oxford-Mahosot Hospital Wellcome Trust Research Unit (Other); Building Resources Across Communities (BRAC), Bangladesh (Unknown); Mahidol Oxford Tropical Medicine Research Unit (Other); Action for Health Development (AHEAD) (Unknown)
Responsible Party: Sponsor
Other Study IDs: BAC20001
Record Dates: First submitted 2020-07-09; First posted 2020-07-20 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Febrile Illness
Keywords: Febrile Illness; Incidence; Causes; Outcomes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Dried blood spots (DBS)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with febrile illness: Participants from approximately 650 villages, with a target number of 100,000 episodes of febrile illness, will be enrolled into this study.

SUMMARY:
The study will collect information to understand the causes and outcomes of febrile illness in rural areas in countries across South and Southeast Asia ( including Cambodia, Laos, Myanmar and Bangladesh). The findings will be used to identify new tests and treatments that can improve the management of febrile patients in the future.

This study is funded by the UK Wellcome Trust. The grant reference number is 215604/Z/19/Z

DETAILED DESCRIPTION:
This study aims to better understand and quantify the burden of febrile illness, the aetiological causes and the manner in which it affects the people living in rural areas in South and Southeast Asia, all on a scale which has not been attempted before. The SEACTN RFI project will collect information to help better understand and predict these outcomes based on a multitude of factors, which will form the basis for interventions within the network in the future. Determining the incidence, causes and outcomes of febrile illness in these settings will be done through two work packages. The first of these, Work Package A (WP-A), the subject of this study, will be carried out at the community level, primarily by engaging village health worker (VHWs) and low-level Health Centres (HCs) which serve the communities to recruit patients presenting with a febrile illness. These patients will be assessed for presenting symptoms and followed up for clinical outcomes. Collection of specimen for diagnostic investigations in these settings is challenging. Currently, mRDTs are conducted by VHWs and HCs in these networks, therefore by using the same process, but also applying blood to filter paper and allowing it to dry (DBS), investigators will test for certain other pathogens, which will increase the aetiological yield.

ELIGIBILITY:
Inclusion Criteria:

* Documented fever (≥ 37.5°C axillary), hypothermia (< 35.5°C) and/or history of fever in the last 24 hours.
* Willingness and ability to comply with study protocol for the study duration.
* Written informed consent given to participate in the trial.

Exclusion Criteria:

* Currently enrolled in the study
* Accident or trauma is the cause for presentation
* Presentation ≤ 3 days after routine immunisations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with an acute febrile illness of all ages presenting to village health workers (VHWs) or peripheral health facilities.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2021-08-04 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Local incidence of febrile illness | From Months 0 to 24
  The incidence per year that an individual seeks care for a febrile illness with the village health workers or local health facility, at the village level.
Overall incidence of febrile illness | From Months 0 to 24
  The incidence per year that an individual seeks care for a febrile illness with the village health workers or local health facility, at the regional level. These estimates will later be triangulated with and extrapolated from using health seeking behavior surveys for an estimate of the total incidence of febrile illness.
Mortality | Within approximately 1 month of first presentation to the village health worker or health facility
  Case fatality rates in febrile illness
Morbidity | Over 1 month after first presentation
  Duration of illness in patients presenting with a fever to the village health worker or health facility.

SECONDARY OUTCOMES:
Prevalence of pathogens in febrile patients | Samples collected over approximately 24 months
  Pathogens will be detected in patients presenting over a 24 month period using point of care tests and diagnostic assays on acute and convalescent dried blood spots.
The correlation between host biomarker concentrations, aetiological diagnoses and clinical outcomes. | Samples collected over approximately 24 months
  The area under the curve, sensitivity and specificity of host biomarkers to identify bacterial infections and to predict severe outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Yoel Lubell, Prof, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (7):
- Building Resources Across Communities (BRAC), Dhaka, Bangladesh
- Medical Action Myanmar (MAM), Yangon, Burma
- Action for Health Development (AHEAD), Battambang, Cambodia
- Lao-Oxford-Mahosot Hospital-Wellcome Trust Research Unit (LOMWRU), Vientiane, Vientiane Prefecture, Laos
- Thailand (3):
  - Mahidol VivaResearch Unit, Faculty of Tropical Medicine, Mahidol University (MVRU), Ratchathewi, Bangkok
  - Shoklo Malaria Research Unit (SMRU), Mae Sot, Changwat Tak
  - Chiangrai Clinical Research Unit (CCRU), Chiang Rai

IPD SHARING:
Plan to Share IPD: Yes
Data collected for this study will be under the custodianship of MORU. With participant's consent, data from this study may be shared in a de-identified form with other groups or researchers in accordance with the MORU Data Sharing Policy.
Time Frame: After completion of trial activities and reporting
Access Criteria: MORU Data Sharing Policy. (http://www.tropmedres.ac/data-sharing-policy)